CLINICAL TRIAL: NCT02824510
Title: Evaluation of Glycemic Changes and Optimization of Glycemic Control During Exercise in Children With Type 1 Diabetes Under Continuous Subcutaneous Insulin Infusion (CSII) or Multiple Daily Injection Regimen (MDI) (TREAD-DIAB Study)
Brief Title: Evaluation of Glycemic Changes During Exercise in Children With Type 1 Diabetes
Acronym: TREAD-DIAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/18NOV/510
Record Dates: First submitted 2016-06-29; First posted 2016-07-06 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart; Insulin Glargine; Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients under insulin pump therapy. (Active Comparator): Patients under insulin pump therapy. Intervention= 2 treadmill exercises to evaluate the efficacy of algorithmic changes in insulin therapy (insulin aspart).
  Interventions: Other: Algorithmic changes in insulin therapy.; Other: Treadmill exercises; Drug: Insulin aspart, glargine and detemir
- Patients under MDI. (Active Comparator): Patients under multiple daily injection regimen. Intervention= 2 treadmill exercises to evaluate the efficacy of algorithmic changes in insulin therapy (insulin aspart and glargine or detemir).
  Interventions: Other: Algorithmic changes in insulin therapy.; Other: Treadmill exercises

INTERVENTIONS:
Other: Algorithmic changes in insulin therapy. — Based on SG evolution in first treadmill test, algorithms will evaluate the modifications in insulin therapy required to normalize SG during the second treadmill test.
Other: Treadmill exercises — 25 min treadmill exercise at 60% of maximal heart rate estimated for age
Drug: Insulin aspart, glargine and detemir
  Arms: Patients under insulin pump therapy.

SUMMARY:
The objectives of the study are: 1) to evaluate the effects of moderate exercise on SG evolution without insulin dose modification in patients with T1D under continuous subcutaneous insulin infusion (CSII) and multiple daily injection (MDI) therapy, and compare differences between these 2 groups; 2) to evaluate the impact of insulin dose modification (bolus, basal, reduction or increase, based on SG evolution profile obtained after first exercise) before and/or during moderate exercise on T1D children under CSII and MDI regimen, and compare differences between these 2 groups.

DETAILED DESCRIPTION:
Intervention and procedures:

a) The patients will first be assigned to standardized moderate-to-vigorous exercise for SG determination; b) similar exercise will then be repeated with preemptive adaptation of insulin dose (tailored on SG evolution during first exercise) for determination of potential influences on SG evolution.

Intervention Plan:

* At first visit (day [>18h] before exercise): setting of a Continuous Glucose Monitoring System
* At second visit: moderate-to-vigorous exercise with treadmill.
* At third visit (2 days after exercise): removal of CGMS
* At fourth visit (day [>18h] before fifth visit): setting of a Continuous Glucose Monitoring System
* At fifth visit: moderate exercise with treadmill, and insulin dose modification (basal rate, bolus, reduction, increase)
* At sixth visit (2 days after exercise): removal of CGMS
* Total number of visits: 6
* The exercises will be performed between 1 and 2 hours after breakfast or after lunch; the second exercise will be performed ≥2 weeks after the first exercise.

Controls:

* Moderate exercise with and without modification of insulin dose in MDI patients (by comparison with CSII patients). MDI patients will be matched to CSII patients according to gender, age, BMI (±0.5 z-score) and HbA1C levels (±1%) to exclude any bias in patient allocation.
* Moderate exercise without modification of insulin dose at first visit (by comparison with modification of insulin dose).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T1D (according to the ISPAD 2011 guidelines)
* T1D outside of partial remission phase (defined according to the IDAA1C definition [Diabetes Care 2007], being equal to A1C (%) + [4 x insulin dose (units per kilogram per 24 h)] and at least > 2 years after T1D diagnosis (defined as the first day of insulin therapy)

Exclusion Criteria:

* Non-type 1 diabetes
* Severe neonatal asphyxia (defined as Apgar score 3 or less after 5 min), children born small for gestational age, chronic systemic disease, active malignancy, hypothyroidism, hypopituitarism, developmental delay, bladder dysfunction, obesity, carnitine deficiency, β-oxidation defect, cardiac malformations, dysrhythmia
* Intake of drugs interfering with insulin sensitivity (e.g. corticosteroids, GH).
* HbA1C >9.5% at the time of enrollment in the study.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2014-08; Primary Completion 2016-09 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Subcutaneous glucose evolution | 12 months
  Subcutaneous glucose evolution after completion of 2 exercise tests

CONTACTS AND LOCATIONS:
Overall Officials: Philippe A Lysy, MD PhD, Principal Investigator — Cliniques Universitaires Saint Luc, Belgium
Locations (1):
- Pediatric Endocrinology, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Moniotte S, Owen M, Barrea T, Robert A, Lysy PA. Outcomes of algorithm-based modifications of insulinotherapy during exercise in MDI vs insulin pump-treated children with type 1 diabetes: Results from the TREAD-DIAB study. Pediatr Diabetes. 2017 Dec;18(8):925-933. doi: 10.1111/pedi.12509. Epub 2017 Mar 2. PMID 28251726